CLINICAL TRIAL: NCT01668537
Title: A Randomized, Double-blind, Multicenter Phase II Trial to Compare the Immunogenicity and Safety of a Liquid-frozen and a Freeze-dried Formulation of IMVAMUNE® (MVA-BN®) Smallpox Vaccine in Vaccinia-naïve Healthy Subjects
Brief Title: A Phase II Trial to Compare a Liquid-frozen and a Freeze-dried Formulation of IMVAMUNE (MVA-BN®) Smallpox Vaccine in Vaccinia-naïve Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: POX-MVA-027
Record Dates: First submitted 2012-08-14; First posted 2012-08-20 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): LF formulation of IMVAMUNE® 2 doses of 1 x 10E8 TCID50, s.c., 4 weeks apart
  Interventions: Biological: LF formulation of IMVAMUNE®
- Group 2 (Experimental): FD formulation of IMVAMUNE® 2 doses of 1 x 10E8 TCID50, s.c., 4 weeks apart
  Interventions: Biological: FD formulation of IMVAMUNE®

INTERVENTIONS:
Biological: LF formulation of IMVAMUNE®
  Arms: Group 1
Biological: FD formulation of IMVAMUNE®
  Arms: Group 2

SUMMARY:
A randomized, double-blind, multicenter Phase II trial to compare the immunogenicity and safety of a liquid-frozen and a freeze-dried formulation of IMVAMUNE (MVA-BN®) smallpox vaccine in vaccinia-naïve healthy subjects

ELIGIBILITY:
Inclusion criteria

1. Male and female subjects, 18-55 years of age
2. The subject has read, signed and dated informed consent form, having been advised of the risks and benefits of the trial in a language understood by the subject and prior to performance of any trial specific procedures and has signed the Health Insurance Portability and Accountability Act (HIPAA) authorization form
3. Body Mass Index (BMI) ≥ 18.5 and < 35
4. Women of childbearing potential (WOCBP) must have used an acceptable method of contraception for 30 days prior to the first vaccination, must agree to use an acceptable method of contraception during the trial, and must avoid becoming pregnant for at least 28 days after the last vaccination. A woman is considered of childbearing potential unless post-menopausal or with a history of hysterectomy. (Acceptable contraception methods are restricted to abstinence, barrier contraceptives, intrauterine contraceptive devices or licensed hormonal products)
5. WOCBP must have a negative serum pregnancy test at screening (SCR) and a negative urine pregnancy test within 24 hours prior to each vaccination
6. White blood cells ≥ 2500/mm3 and < ULN
7. Absolute neutrophil count (ANC) within normal limits
8. Hemoglobin within normal limits
9. Platelets within normal limits
10. Adequate renal function defined as a calculated Creatinine Clearance (CrCl) > 60 ml/min as estimated by the Cockcroft-Gault equation:

    * For men: (140 - age in years) x (body weight in kg) ÷ (serum creatinine in mg/dl x 72) = CrCl (ml/min)
    * For women: multiply the result by 0.85 = CrCl (ml/min)
11. Adequate hepatic function defined as:

    * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) in the absence of other evidence of significant liver disease
    * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase < 1.5 x ULN
12. Troponin I < 2 x ULN
13. Electrocardiogram (ECG) without clinically significant findings, e.g. any kind of atrioventricular or intraventricular conditions or blocks such as complete left or right bundle branch block, AV node block, QTc or PR prolongation, premature atrial contractions or other atrial arrhythmia, sustained ventricular arrhythmia, two premature ventricular contractions (PVC) in a row, ST elevation consistent with ischemia

Exclusion criteria

1. Typical vaccinia scar
2. Known or suspected history of smallpox vaccination
3. History of vaccination with any poxvirus-based vaccine
4. US Military service before 1991 or after January 2003
5. Pregnant or breast-feeding women
6. Uncontrolled serious infection, i.e. not responding to antimicrobial therapy
7. History of any serious medical condition, which in the opinion of the investigator would compromise the safety of the subject or would limit the subject's ability to complete the trial in the opinion of the investigator
8. History of or active autoimmune disease, persons with vitiligo or thyroid disease taking thyroid hormone replacement are not excluded
9. Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease, diabetes mellitus, moderate to severe kidney impairment
10. History of malignancy, other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure. Subjects with history of skin cancer must not be vaccinated at the previous tumor site
11. History or clinical manifestation of clinically significant and severe hematological, pulmonary, central nervous, cardiovascular or gastrointestinal disorders
12. Clinically significant mental disorder not adequately controlled by medical treatment
13. History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, or any other heart condition under the care of a doctor
14. History of an immediate family member (father, mother, brother, or sister) who has had onset of ischemic heart disease before the age of 50 years
15. Twenty percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's Risk Assessment Tool: http://hin.nhlbi.nih.gov/atpiii/calculator.asp NOTE: This criterion applies only to subjects 20 years of age and older
16. Active or history of chronic alcohol abuse and/or intravenous and/or nasal drug abuse (within the past 6 months)
17. Known allergy to IMVAMUNE® vaccine and its constituents, e.g. tris(hydroxymethyl)-amino methane, including known allergy to egg or aminoglycoside (gentamycin)
18. History of anaphylaxis or severe allergic reaction to any vaccine
19. Acute disease (illness with or without a fever) at the time of enrollment
20. Body Temperature ≥ 100.4°F (38.0°C) at the time of enrollment
21. Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior or after trial vaccination
22. Having received any vaccinations or planned vaccinations with a killed vaccine within 14 days prior or after trial vaccination
23. Chronic systemic administration (defined as more than 14 days) of > 5 mg prednisone (or equivalent)/day or any other immune-modifying drugs during a period starting from three months prior to administration of the vaccine and ending at last physical trial visit (Visit 5)
24. Post organ transplant subjects whether or not receiving chronic immunosuppressive therapy
25. Administration or planned administration of immunoglobulins and/or any blood products during a period starting from three months prior to administration of the vaccine and ending at last physical trial visit (Visit 5)
26. Use of any investigational or non-registered drug or vaccine other than the trial vaccine within 30 days preceding the first dose of the trial vaccine or planned administration of such a drug during the trial period (with the day of the FU call being considered the last day of the trial period).
27. Trial personnel

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 651 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard N Greenberg, MD, Principal Investigator — University of Kentucky
Locations (3):
- United States (3):
  - Miami Research Associates, South Miami, Florida
  - PRA, Lenexa, Kansas
  - University of Kentucky, Lexington, Kentucky

RESULTS

PARTICIPANT FLOW:
Groups:
- LF Formulation: Liquid Frozen (LF) formulation of MVA-BN® 2 doses of 1 x 10E8 TCID50, subcutaneous (s.c.), 4 weeks apart
  LF formulation of MVA-BN®
- FD Formulation: Freeze Dried (FD) formulation of MVA-BN® 2 doses of 1 x 10E8 TCID50, s.c., 4 weeks apart
  FD formulation of MVA-BN®
Period: Overall Study
Arm/Group | LF Formulation | FD Formulation
Started (randomized and vaccinated) | 327 | 324
Completed (active trial phase) | 305 | 314
Not Completed | 22 | 10
Not completed — Request to Discontinue Prematurely | 1 | 1
Not completed — Subject unwilling/unable to comply | 5 | 0
Not completed — Reason Precludes Participation | 1 | 0
Not completed — Lost to Follow-up | 13 | 6
Not completed — Other | 2 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- LF Formulation: Liquid Frozen formulation of MVA-BN® 2 doses of 1 x 10E8 TCID50, s.c., 4 weeks apart
  LF formulation of MVA-BN®
- FD Formulation: Freeze Dried formulation of MVA-BN® 2 doses of 1 x 10E8 TCID50, s.c., 4 weeks apart
  FD formulation of MVA-BN®
- Total: Total of all reporting groups
Arm/Group | LF Formulation | FD Formulation | Total
Number analyzed (Participants) | 327 | 324 | 651
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (6.36) | 27.6 (6.21) | 27.7 (6.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 170 | 348
  Male | 149 | 154 | 303
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 95 | 95 | 190
  Not Hispanic or Latino | 232 | 229 | 461
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 78 | 67 | 145
  White | 239 | 247 | 486
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 327 | 324 | 651

OUTCOME MEASURES:

1. Primary Outcome: ELISA GMT
Description: Geometric Mean Titers (GMT) based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Titers below the detection limit are included with a value of '1'
Time Frame: Week 6
Population: Per Protocol Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 297 | 306
Titer | 875.1 [801.3 to 955.7] | 1099.6 [1014.8 to 1191.6]
Statistical Analysis 1: Comparison: LF Formulation vs FD Formulation; Test type: Non-Inferiority — The non-inferiority margin to show that the FD formulation is non-inferior to the LF formulation in terms of ELISA GMTs at the peak visit (Week 6) was predefined as '1.5' for the GMT ratio (LF/FD). Non-inferiority is demonstrated if the upper 95% CI of the GMT ratio (LF/FD) is entirely below 1.5; GMT ratio (LF/FD) = 0.796, 95% CI 2-sided [0.707 to 0.896]

2. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Occurrence, relationship to the trial vaccine and intensity of any Serious Adverse Event (SAE).
Time Frame: up to 32 weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 327 | 324
Participants
  SAE | 5 | 2
  SAE related to vaccine | 0 | 0
  SAE Grade >=3 | 3 | 1

3. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI)
Description: Occurrence, relationship to the trial vaccine and intensity of any Adverse Event of Special Interest (AESI). AESIs were defined as any cardiac symptoms and ECG changes determined to be clinically significant or cardiac enzyme troponin I elevated above 2 x the Upper Limit of Normal
Time Frame: up to 32 weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 327 | 324
Participants
  AESI | 1 | 4
  Drug-related AESI | 0 | 0
  AESI Grade >=3 | 0 | 0

4. Secondary Outcome: Number of Participants With Related Grade >=3 Adverse Events
Description: Occurrence of any Grade >=3 Adverse Events related to the trial vaccine.
Time Frame: within 29 days after vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 327 | 324
Participants | 0 | 1

5. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: Occurrence, relationship to the trial vaccine and intensity of unsolicited treatment-emergent AEs (TEAEs).
Time Frame: within 29 days after vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 327 | 324
Participants
  TEAE | 313 | 310
  Drug-Related TEAE | 207 | 207
  TEAE Grade >=3 | 6 | 5
  Drug-Related TEAE Grade >=3 | 0 | 1

6. Secondary Outcome: Number of Participants With Solicited Local Averse Events
Description: Occurrence and intensity of solicited local AEs (redness, swelling, induration, pruritus and pain) during the 8-day period (day of vaccination and the following 7 days) after any vaccination. Events were graded by intensity (1 = mild, 2 = moderate, 3 = severe).
Time Frame: 8 days after any vaccination
Population: Subjects of the Full Analysis Set with at least one completed diary card
Measure: Number; unit: participants
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 322 | 321
participants
  Injection site pain : All | 274 | 290
  Injection site pain : Grade >=2 | 138 | 167
  Injection site pain : Grade =3 | 22 | 35
  Injection site erythema : All | 247 | 255
  Injection site erythema : Grade >=2 | 140 | 181
  Injection site erythema : Grade =3 | 16 | 47
  Injection site swelling : All | 210 | 223
  Injection site swelling : Grade >=2 | 94 | 125
  Injection site swelling : Grade =3 | 10 | 23
  Injection site induration : All | 211 | 213
  Injection site induration : Grade >=2 | 73 | 96
  Injection site induration : Grade =3 | 5 | 6
  Injection site pruritus : All | 177 | 189
  Injection site pruritus : Grade >=2 | 38 | 47
  Injection site pruritus : Grade =3 | 7 | 11

7. Secondary Outcome: Number of Participants With Solicited General Adverse Events
Description: Occurrence, intensity and relationship to the trial vaccines of solicited general AEs (pyrexia, headache, myalgia, nausea, fatigue and chills) during the 8-day period (day of vaccination and the following 7 days) after any vaccination. Events were graded by intensity (1 = mild, 2 = moderate, 3 = severe).
Time Frame: within 8 days after any vaccination
Population: Subjects of the Full Analysis Set with at least one completed diary card
Measure: Number; unit: participants
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 322 | 321
participants
  Body Temperature increased : All | 23 | 33
  Body Temperature increased : Grade >=2 | 7 | 8
  Body Temperature increased : Grade =3 | 3 | 2
  Body Temperature increased : Related | 22 | 30
  Body Temperature increased : Related Grade =3 | 3 | 2
  Headache : All | 125 | 112
  Headache : Grade >=2 | 37 | 27
  Headache : Grade =3 | 8 | 7
  Headache : Related | 110 | 94
  Headache : Related Grade =3 | 6 | 6
  Myalgia : All | 68 | 59
  Myalgia : Grade >=2 | 24 | 18
  Myalgia : Grade =3 | 1 | 5
  Myalgia : Related | 59 | 47
  Myalgia : Related Grade =3 | 1 | 3
  Chills : All | 38 | 35
  Chills : Grade >=2 | 14 | 10
  Chills : Grade =3 | 2 | 5
  Chills : Related | 34 | 33
  Chills : Related Grade =3 | 2 | 4
  Nausea : All | 57 | 51
  Nausea : Grade >=2 | 19 | 18
  Nausea : Grade =3 | 4 | 2
  Nausea : Related | 53 | 44
  Nausea : Related Grade =3 | 4 | 2
  Fatigue : All | 113 | 102
  Fatigue : Grade >=2 | 39 | 39
  Fatigue : Grade =3 | 15 | 9
  Fatigue : Related | 106 | 95
  Fatigue : Related Grade =3 | 14 | 9

8. Secondary Outcome: ELISA GMTs
Description: Geometric Mean Titers (GMT) at all immunogenicity sampling time points based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). For the calculation of GMTs all measurements are included as they provide meaningful information even if below the detection limit (DL). Disregarding these measurements would highly bias the reported GMTs. We imputed values <DL as a value of '1' and the GMT and corresponding 95% confidence intervals were calculated.
Time Frame: within 8 weeks
Population: Per Protocol Analysis Set. Number Analyzed refers to the number of participants with measurements at the respective sampling time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 297 | 306
Titer
  Week 0 | 1.1 [1.0 to 1.2] | 1.1 [1.0 to 1.2]
  Week 2 | 56.0 [44.8 to 69.9] | 90.4 [75.9 to 107.7]
  Week 4: number analyzed (Participants) | 297 | 305
  Week 4 | 89.6 [75.0 to 107.0] | 131.3 [115.8 to 148.9]
  Week 6 | 875.1 [801.3 to 955.7] | 1099.6 [1014.8 to 1191.6]
  Week 8 | 546.4 [499.4 to 597.8] | 689.0 [635.2 to 747.4]

9. Secondary Outcome: PRNT GMT
Description: Geometric Mean Titers (GMT) based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Titers below the detection limit are included with a value of '1'
Time Frame: Week 6
Population: Per Protocol Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 297 | 306
Titer | 81.8 [73.0 to 91.6] | 101.2 [91.0 to 112.5]

10. Secondary Outcome: PRNT GMTs
Description: Geometric Mean Titers (GMT) at all immunogenicity sampling time points based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). For the calculation of GMTs all measurements are included as they provide meaningful information even if below the detection limit (DL). Disregarding these measurements would highly bias the reported GMTs. We imputed values <DL as a value of '1' and the GMT and corresponding 95% confidence intervals were calculated.
Time Frame: within 8 weeks
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 297 | 306
Titer
  Week 0 | 1.1 [1.0 to 1.1] | 1.0 [1.0 to 1.1]
  Week 2 | 7.1 [6.0 to 8.6] | 10.4 [8.7 to 12.3]
  Week 4: number analyzed (Participants) | 297 | 305
  Week 4 | 9.3 [7.9 to 11.1] | 12.5 [10.6 to 14.7]
  Week 6 | 81.8 [73.0 to 91.6] | 101.2 [91.0 to 112.5]
  Week 8 | 59.7 [54.0 to 66.0] | 76.1 [69.6 to 83.2]

11. Secondary Outcome: Percentage of Participants With Seroconversion by ELISA
Description: Seroconversion rate based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (50) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects.
Time Frame: Week 6
Population: Per Protocol Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 297 | 306
percentage of subjects | 100.0 | 100.0

12. Secondary Outcome: Percentage of Participants With Seroconversion by ELISA
Description: Seroconversion rates at all post-baseline immunogenicity sampling time points based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (50) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: within 8 weeks
Population: as for outcome 8
Measure: Number; unit: percentage of subjects
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 297 | 306
percentage of subjects
  Week 2 | 83.5 | 91.5
  Week 4: number analyzed (Participants) | 297 | 305
  Week 4 | 91.9 | 97.0
  Week 6 | 100.0 | 100.0
  Week 8 | 100.0 | 100.0

13. Secondary Outcome: Percentage of Participants With Seroconversion by PRNT
Description: Seroconversion rate based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (2) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects.
Time Frame: Week 6
Population: Per Protocol Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 297 | 306
percentage of subjects | 99.0 | 100.0

14. Secondary Outcome: Percentage of Participants With Seroconversion by PRNT
Description: Seroconversion rates at all post-baseline immunogenicity sampling time points based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Seroconversion is defined as the appearance of antibody titers ≥ detection limit (2) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: within 8 weeks
Population: as for outcome 8
Measure: Number; unit: percentage of subjects
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 297 | 306
percentage of subjects
  Week 2 | 80.1 | 87.3
  Week 4: number analyzed (Participants) | 297 | 305
  Week 4 | 84.8 | 91.5
  Week 6 | 99.0 | 100.0
  Week 8 | 100.0 | 99.7

15. Secondary Outcome: ELISPOT Magnitudes of Response
Description: Magnitudes of response of IFNγ producing T-cells measured by vaccinica-specific ELISPOT. Spot Forming Units below the detection limit are included as a value of '1'.
Time Frame: within 8 weeks
Population: ELISPOT Analysis Set
Measure: Median (95% Confidence Interval); unit: Spot Forming Units
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 101 | 94
Spot Forming Units
  Week 0 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Week 2 | 393.0 [318.0 to 506.0] | 581.5 [416.0 to 718.0]
  Week 4 | 88.0 [70.0 to 107.0] | 133.0 [100.0 to 170.0]
  Week 6 | 235.0 [185.0 to 343.0] | 315.0 [232.0 to 412.0]
  Week 8 | 145.5 [115.0 to 174.0] | 240.0 [146.0 to 284.0]

16. Secondary Outcome: Percentage of Participants With Response by ELISPOT
Description: Response rates regarding IFNγ producing T-cells measured by vaccinia-specific ELISPOT. A response to the vaccine was defined as either the appearance of a positive signal for participants without a positive signal at Baseline or an increase by a factor of at least 1.7 of the SFU/1 x 10E6 PBMC compared to the Baseline SFU/1 x 10E6 PBMC for participants with a positive signal at Baseline.
Time Frame: within 8 weeks
Population: ELISPOT Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 101 | 94
percentage of subjects
  Week 2 | 95.0 | 97.9
  Week 4 | 66.0 | 80.2
  Week 6 | 88.0 | 94.4
  Week 8 | 84.0 | 92.3

17. Secondary Outcome: Percentage of Responders by ELISPOT
Description: Responder rate measured by vaccinia specific ELISPOT. A participant was defined as a responder to the vaccine determined by ELISPOT if the participant had at least 1 post-baseline visit determined to be a response. A response to the vaccine was defined as either the appearance of a positive signal for participants without a positive signal at Baseline or an increase by a factor of at least 1.7 of the SFU/1 x 10E6 PBMC compared to the Baseline SFU/1 x 10E6 PBMC for participants with a positive signal at Baseline.
Time Frame: within 8 weeks
Population: ELISPOT Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 101 | 94
percentage of subjects | 100 | 100

18. Secondary Outcome: Correlation ELISA vs PRNT Titers
Description: Pearson Correlation Coefficient between the ELISA titers and the PRNT titers at weeks 4, 6 and 8 based on the log10 transformed titer values
Time Frame: within 8 weeks
Population: Per Protocol Analysis Set
Measure: Number (95% Confidence Interval); unit: Pearson Correlation Coefficient
Arm/Group | LF Formulation | FD Formulation
Number analyzed (Participants) | 297 | 306
Pearson Correlation Coefficient
  Week 4: number analyzed (Participants) | 297 | 305
  Week 4 | 0.597 [0.518 to 0.665] | 0.492 [0.401 to 0.572]
  Week 6 | 0.646 [0.574 to 0.708] | 0.553 [0.470 to 0.627]
  Week 8 | 0.567 [0.484 to 0.640] | 0.565 [0.484 to 0.637]

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | LF Formulation | FD Formulation
All-Cause Mortality (participants affected / at risk) | 0/327 | 0/324
Serious Adverse Events (participants affected / at risk) | 5/327 | 2/324
Other Adverse Events (participants affected / at risk) | 115/327 | 114/324
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LF Formulation (N=327) | FD Formulation (N=324)
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LF Formulation (N=327) | FD Formulation (N=324)
Injection site induration (General disorders) | 77 | 74
Injection site hemorrhage (General disorders) | 2 | 17
Injection site pain (General disorders) | 6 | 7
Injection site discoloration (General disorders) | 5 | 9
Injection site hematoma (General disorders) | 5 | 5
Fatigue (General disorders) | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 16 | 19
Viral upper respiratory tract infection (Infections and infestations) | 12 | 8
Headache (Nervous system disorders) | 8 | 5
Vomiting (Gastrointestinal disorders) | 4 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes